CLINICAL TRIAL: NCT01360372
Title: The Effect Of Methylnaltrexone (Relistor™) on Gut Motility and Tolerance to Tube Feeding in Patients Treated With Opiate Therapy
Brief Title: Effect of Methylnaltrexone (Relistor) on Digestion and Tolerance to Tube Feeding in Patients Treated With Opiates
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No eligible subjects identified
Sponsor: Drexel University (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Michael Sherman, MD PI, Drexel University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Drexel18538
Record Dates: First submitted 2011-03-16; First posted 2011-05-25 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Tube Feeding
Keywords: Hydrogen breath test value and gastric residual volume measurements; Tube feeding tolerance while taking a stable dose of opiate
MeSH Terms: interventions — methylnaltrexone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylnaltrexone (Active Comparator)
  Interventions: Drug: Methylnaltrexone
- saline placebo injection (Placebo Comparator)
  Interventions: Drug: Saline injection

INTERVENTIONS:
Drug: Methylnaltrexone — Methylnaltrexone 8 mg IV for subjects 38 to 62 kg body weight, Methylnaltrexone12 mg IV for subjects 62.1 to 114 kg body weight
  Arms: Methylnaltrexone
Drug: Saline injection — Saline 0.4 to 0.8 ml injection
  Arms: saline placebo injection

SUMMARY:
It is hypothesized that using methylnaltrexone in addition to pain killer narcotics (opiates) in patients will result in increased tube feeding rates with more frequent nutrition at goal calorie rate.

DETAILED DESCRIPTION:
Tube feeding rates and tube feeding residual volumes will be measured and followed blinded to the treatment arm (methylnaltrexone vs. placebo) to evaluate if patients (who prior to study entry did not tolerate goal rates tube feeds) can get closer to tube feeding goal with the treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Inadequate tube feeding rate of greater than equal to 40% below goal rate.
* Prescribed opiate therapy for pain or sedation, stable dose for minimum 48 hours
* Stable dose or no dose laxative for minimum 72 hours

Exclusion Criteria:

* Unstable Hemodynamics (eg. vasopressor medication)
* Pregnancy
* End stage Renal Disease on Dialysis
* Plan to wean opiates in next 48 hours
* Known or suspected mechanical gastrointestinal obstruction
* Initial expired hydrogen breath level greater than 20

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Hydrogen breath test measure of bowel transit | 2 days
  On day 1 Hydrogen Breath Test (HBT) measures will occur 30 minutes before test meal, immediately after test meal every 15 minutes until a rise of 5ppm is detected or until 4 hours have passed. On day 2 Hydrogen Breath test measures will occur 30 minutes before test meal, immediately after test meal and every 15 minutes until a rise of 5ppm is detected or until 4 hours have passed.

SECONDARY OUTCOMES:
Gastric residual volume measurement | 3 days
  Gastric residual volumes will be measured at baseline study entry and then every 4 hours throughout the study until 24 hours post study drug administration.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Cancer Treatment Center of America, Philadelphia, Pennsylvania